CLINICAL TRIAL: NCT05107700
Title: The Impact of Hypoxia on Patients With Precapillary Pulmonary Hypertension and Treatment of Adverse Effects
Brief Title: Altitude Related Adverse Health Effects (ARAHE) in Patients With Precapillary Pulmonary Hypertension During 30h Exposure to 2500m
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: OVERALP II A
Record Dates: First submitted 2021-10-12; First posted 2021-11-04 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: High Altitude Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary edema of mountaineers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Start with: Stay at altitude 2500 m above sea level (high altitude) (Experimental): Patients with precapillary pulmonary hypertension stay a sojourn of 30 h at 2500 m.
  Interventions: Procedure: Stay at altitude 2500 m above sea level (high altitude); Procedure: Stay at altitude 470 m above sea level (low altitude)
- Start with: Stay at altitude 470 m above sea level (low altitude) (Placebo Comparator): Patients with precapillary pulmonary hypertension stay a sojourn of 30 h at 470 m as comparator.
  Interventions: Procedure: Stay at altitude 2500 m above sea level (high altitude); Procedure: Stay at altitude 470 m above sea level (low altitude)

INTERVENTIONS:
Procedure: Stay at altitude 2500 m above sea level (high altitude) — Patients with precapillary pulmonary hypertension stay a sojourn of 30 h at 2500 m.
Procedure: Stay at altitude 470 m above sea level (low altitude) — Patients with precapillary pulmonary hypertension stay a sojourn of 30 h at 470 m.

SUMMARY:
The interest of journeys to high altitude regions for recreational or professional purposes is increasing, also among potentially vulnerable groups including patients with chronic cardiopulmonary diseases such as pulmonary hypertension (PH). In Switzerland and many other regions worldwide, many settlements and alpine resorts are at altitudes above 1500m and alpine tourism is an important social and economic sector. However, the hypoxic environment at altitude may induce altitude related adverse health effects (ARAHE), including hypoxemia, symptoms of acute mountain sickness (AMS), reduces exercise capacity and increases the pulmonary arterial pressure, which is of particular relevance for patients with chronic hypoxemic respiratory diseases including PH.

On the other hand, advances in disease-targeted medical combination therapies renders PH to the chronic disease groups with many patients surviving for many years with a relatively good quality of live, exercise capacity and low symptom burden. However, data on ARAHE and the exercise capacity of patients with pre-existing PH at altitude is scarce, so that current expert-based guidelines discourage altitude travel for patients with PH. However, we previously showed that the majority of stable PH-patients tolerates normobaric hypoxia or a short trip to 2500m well.

With this project we aim to get profound clinical and pathophysiological insights into the effects of the hypobaric hypoxic environment at altitude during an overnight stay up to 30 hours on the incidence of ARAHE needing oxygen therapy, exercise capacity, pulmonary hemodynamics and sleep in patients with precapillary PH.

We hope that this new valuable data will provide a basis to better counsel PH-patients for potential risk of altitude sojourns.

DETAILED DESCRIPTION:
Background:

Precapillary PH is defined by right heart catheterization as mean PAP (mPAP) >20 mmHg, pulmonary artery wedge pressure (PAWP) ⩽15 mmHg along with a pulmonary vascular resistance (PVR) ⩾3 wood units (WU). PH is classified into five major groups according to the clinical presentation and response to vasodilator therapies. In the absence of predominant lung disease, the major precapillary PH forms are pulmonary arterial and chronic thromboembolic PH that are the main pulmonary vascular diseases and hereafter summarized as PH.

The leading symptom in PH is dyspnoea on exertion, impaired exercise performance, daily activity and quality of life.With progression of the disease, worsening hemodynamics may lead to gas exchange disturbances associated with hypoxemia, particularly during exercise and sleep. For a long time, the occurrence of PH was associated with a dismal prognosis progressively leading to right heart failure and death within months to a few years. Although PH is still incurable, recent therapeutic advances including medical or interventional therapies have improved the life expectancy, physical performance and quality of life of PH-patients and many patients seen in our daily practice wish to near-normally participate in professional work and recreational activities.

Globally, leisure time and professional activities at high altitude become increasingly popular exposing millions of people to hypobaric hypoxia annually. The alpine tourism in Europe and in other regions worldwide has a long lasting tradition and a relevant number of people have chosen their resident above 1500m above sea level.

Travel to high altitude and altitude-related adverse health effects (ARAHE):

Many Swiss villages and tourist resorts are located at altitudes between 1000 - 2500 m. In America, Asia and Africa, even large settlements are located at these or even higher altitudes and it is estimated that more than 50 million people permanently live above 2500 m. Accordingly, worldwide, millions of people travel regularly to mountain areas for business or recreation and expose themselves to hypobaric hypoxia during days to weeks or even longer. In addition, traveling by airplane, which has become extremely popular, further increased the number of people that are exposed to a hypoxic environment, as the minimally allowed cabin pressure in commercial air travel is equivalent to 2430 m (8000 ft) of altitude and this is often reached in intercontinental flights.

In healthy individuals, altitude exposure acutely induces hyperventilation by hypoxic chemoreceptor stimulation. This mitigates hypoxemia but promotes sleep disturbing high-altitude periodic breathing. About 50% of lowlanders ascending rapidly to >3000 m suffer from acute mountain sickness (AMS) causing headache, loss of appetite, weakness, fatigue and general discomfort. If AMS is not treated by descent, oxygen or medication, it may progress to life-threatening high altitude cerebral oedema. Furthermore, hypoxic pulmonary vasoconstriction (HPV) leads to an elevated PAP at altitude. In 2-4% of mountaineers climbing to 4559 m, excessive PAP-increase triggers high altitude pulmonary edema (HAPE), a non-cardiogenic pulmonary oedema associated with profound, potentially life-threatening hypoxemia, which is treated by oxygen therapy and may be prevented by phosphodiesterase type-5 inhibitor (PDE5i) administration or dexamethasone.

Contribution of this project to the gap in knowledge of the effects of hypoxia in PH:

The proposed trials will provide novel, robust data on the clinical and pathophysiological effects of exposure to a hypoxic environment in patients with PAH/CTEPH. This study will evaluate for the first time safety and tolerability of altitude exposure including an overnight stay in PH-patients and the effect of supplemental oxygen to reverse ARAHE. Close monitoring of patients including during exercise and sleep will provide insight into hypoxia-induced physiological mechanisms and the time course of altitude adaptation. Due to the special geographical location of Switzerland, we have the unique opportunity to study the response to hypobaric hypoxia in patients with PH in excellently suitable and safe settings in the nearby mountains and provide this important data to the scientific community worldwide for the benefit of many PH-patients and their advising caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* PH class I (PAH) or IV (CTEPH) diagnosed according to guidelines: mean pulmonary artery pressure >20 mmHg, pulmonary vascular resistance ≥3 wood units, pulmonary arterial wedge pressure ≤15 mmHg during baseline measures at the diagnostic right-heart catheterization

Exclusion Criteria:

* Resting partial pressure of oxygen <8 kilopascal at Zurich at 490 m low altitude
* Exposure to an altitude >1000 m for ≥3 nights during the last 2 weeks before the study
* Inability to follow the procedures of the study
* Other clinically significant concomitant end-stage disease (e.g., renal failure, hepatic dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Incidence of altitude-related adverse health effects (ARAHE as defined below) during a sojourn at 2500m, time frame up to 30 h. ARAHE will be defined by any of the following criteria: | 30 hours
  * Acute mountain sickness with a Lake Louise score >4 including headache, or AMSc score ≥0.7
  * severe hypoxemia defined as: resting SpO2 <75% for >15 min or <80% for >30 min; exercise SpO2 <75% for >5 min and/or criteria for stopping exercise according to guidelines
  * intercurrent illness: infection, neurologic, impairment, other new diseases/accidents, requiring medical treatment other than simple measures such as paracetamol
  * chest pain and/or ECG signs of cardiac ischemia, syncope, tachy- or bradyarrhythmia, severe hyper- or hypotension accompanied by symptoms
  * dyspnoea at rest and/or any discomfort requiring treatment and/or leading to the wish of a patient to return to low altitude or withdraw from the study

SECONDARY OUTCOMES:
Components of altitude-related adverse health effects | 30 hours
  Incidence of individual components of altitude-related adverse health effects
Severity of symptoms | 30 hours
  Severity of symptoms of acute mountain sickness at 2500 m of high altitude measured by the Lake louise score (LLS) (or Acute Mountain Sickness c questionnaire)
Difference in pulmonary artery pressure | 30 hours
  Difference in pulmonary artery pressure assessed by the transtricuspid pressure gradient at rest by echocardiography at high vs. low altitude
Difference in pulmonary vascular resistance assessed | 30 hours
  Difference in pulmonary vascular resistance assessed by the transtricuspid pressure gradient at rest by echocardiography at high vs. low altitude
Difference in right ventricular function | 30 hours
  Difference in right ventricular function impairment by echocardiography at high vs. low altitude
Resting electrocardiography | 30 hours
  Prevalence of abnormal resting electrocardiographies (ECG) at high altitude vs. low altitude
Exercise electrocardiography | 30 hours
  Prevalence of abnormal exercise electrocardiographies (ECG) at high altitude vs. low altitude
Blood pressure | 30 hours
  Difference in blood pressure at high vs. low altitude
Heart-rate variability | 30 hours
  Difference in heart-rate variability at high vs. low altitude

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Muller J, Mayer L, Schneider SR, Bauer M, Furian M, Bloch KE, Schwarz EI, Lichtblau M, Silvia U. Pulmonary haemodynamics and right heart function during exercise at high versus low altitude in patients with pulmonary vascular disease: a randomised crossover trial. Heart. 2025 Dec 11;112(1):28-36. doi: 10.1136/heartjnl-2024-325605. PMID 40404280